CLINICAL TRIAL: NCT03356145
Title: 12 Versus 20 mL Paracervical Block for Pain-Control During Cervical Preparation for Dilation and Evacuation: A Single-Blinded Randomized Controlled Trial
Brief Title: 12 Versus 20 mL PCB for D&E Cervical Prep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-43789
Record Dates: First submitted 2017-11-20; First posted 2017-11-29 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pain
Keywords: paracervical block; abortion; dilation and evacuation; cervical preparation
MeSH Terms: conditions — Pain; Dilatation, Pathologic | interventions — Anesthesia, Obstetrical

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two study arms via computer-generated block randomization using REDCap software.
Who Masked: Participant
Masking Description: The provider and staff will be aware of arm allocation, but participants will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 12 mL arm (Experimental): Intervention:
  * Syringe loaded with 12 mL of 1% lidocaine (120 mg); 22-gauge spinal needle
  * 2 mL injected at the tenaculum site, either 6 or 12 o'clock superficially into the cervix
  * The tenaculum is immediately placed at the previously injected site
  * The remaining 10 mL are slowly injected into the cervicovaginal junction in two equal aliquots at 4 and 8 o'clock; the injection is continuous from superficial to deep (3 cm) to superficial (injecting with insertion and withdrawal)
  * No wait time between injection and dilator insertion
  Interventions: Drug: 12 mL paracervical block
- 20 mL arm (Active Comparator): Intervention:
  * Syringe loaded with 20 mL of 1% lidocaine (120 mg); 22-gauge spinal needle
  * 2 mL injected at the tenaculum site, either 6 or 12 o'clock superficially into the cervix
  * The tenaculum is immediately placed at the previously injected site
  * The remaining 18 mL are slowly injected into the cervicovaginal junction in two equal aliquots at 4 and 8 o'clock; the injection is continuous from superficial to deep (3 cm) to superficial (injecting with insertion and withdrawal)
  * No wait time between injection and dilator insertion
  Interventions: Drug: 20 mL paracervical block

INTERVENTIONS:
Drug: 12 mL paracervical block — Injection of 12 mL of lidocaine
  Arms: 12 mL arm
Drug: 20 mL paracervical block — Injection of 20 mL of lidocaine
  Arms: 20 mL arm

SUMMARY:
More research is needed to investigate methods of pain control for cervical preparation for abortion procedures. Women report pain with paracervical block injection as well as with osmotic dilator placement. This study seeks to compare a 12 mL, 2-site 1% plain lidocaine paracervical block for pain control during cervical preparation (osmotic dilator insertion) for Dilation and Evacuation (D&E) to a 20 mL 1% lidocaine 2-site paracervical block.

DETAILED DESCRIPTION:
This is a non-inferiority, single blinded, randomized controlled trial.This study will use a 2-site, 12 mL 1% plain lidocaine injection paracervical block (PCB) technique (2 mL for tenaculum placement, 10 mL for paracervical block) will provide non-inferior pain control compared to a previously established 2-site, 20 mL 1% lidocaine injection PCB (2 mL for tenaculum placement, 18 mL for paracervical block) when administered for dilation pain control during cervical preparation.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 and older
* Intrauterine pregnancy ≥16 weeks gestation
* English speaking competency
* Willing and able to sign consent forms
* Agree to comply with study procedures

Exclusion Criteria:

* Women less than 18 years of age
* IV conscious sedation
* Known allergy to study medication (lidocaine)
* Any women not meeting inclusion criteria above will be excluded from participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

REFERENCES:
- [Derived] Shaw KA, Lerma K, Hughes T, Hastings C, Fok WK, Blumenthal PD. A Comparison of Paracervical Block Volumes Before Osmotic Dilator Placement: A Randomized Controlled Trial. Obstet Gynecol. 2021 Sep 1;138(3):443-448. doi: 10.1097/AOG.0000000000004485. PMID 34352829

RESULTS

PARTICIPANT FLOW:
Groups:
- 12 mL Arm: Participants receive injection of 12 mL of lidocaine.
- 20 mL Arm: Participants receive injection of 20 mL of lidocaine.
Period: Overall Study
Arm/Group | 12 mL Arm | 20 mL Arm
Started | 48 | 48
Received Allocated Intervention | 45 | 47
Completed | 45 | 47
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Did not meet inclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were allocated to the intervention and for whom primary outcome measure data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | 12 mL Arm | 20 mL Arm | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (7) | 31 (7) | 31 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 91
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 16 | 25
  Not Hispanic or Latino | 36 | 30 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 15 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 46 | 91

OUTCOME MEASURES:

1. Primary Outcome: Pain Immediately Following Dilator Insertion
Description: The primary objective is to determine pain perceived immediately following dilator insertion measured by Visual Analogue Scale (VAS) (0-100mm; 0 being no pain, 100 being worst pain imaginable).
Time Frame: Time of dilator insertion (less than 1 minute to assess pain)
Population: Participants who received the allocated intervention and for whom primary outcome data are available
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 12 mL Arm | 20 mL Arm
Number analyzed (Participants) | 45 | 46
score on a scale | 41 [21 to 58] | 49 [26 to 65]

2. Secondary Outcome: Anticipated Pain Immediately Prior to Dilator Insertion
Description: Pain measured by VAS (0-100mm; 0 being no pain, 100 being worst pain imaginable).
Time Frame: Up to 1 minute to complete survey
Population: Participants who received the allocated intervention and for whom primary outcome data are available
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 12 mL Arm | 20 mL Arm
Number analyzed (Participants) | 45 | 46
score on a scale | 51 [28 to 62] | 58 [43 to 69]

3. Secondary Outcome: Patient Global Satisfaction Score
Description: Global satisfaction (acceptability) of procedure reported by participant, measured by 0-100mm VAS; with anchors at 0 ("worse than expected"), 50 ("what I expected"), and 100 ("better than expected").
Time Frame: Up to 1 minute to complete survey
Population: Participants who received the allocated intervention and for whom primary outcome data are available
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 12 mL Arm | 20 mL Arm
Number analyzed (Participants) | 45 | 46
score on a scale | 70 [39 to 91] | 53 [44 to 87]

4. Secondary Outcome: Total Procedure Time
Description: Defined as time of speculum insertion
Time Frame: Up to 10 minutes
Population: Participants who received the allocated intervention and for whom primary outcome data are available
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 12 mL Arm | 20 mL Arm
Number analyzed (Participants) | 45 | 46
minutes | 5.5 [4.6 to 6.9] | 5.7 [4.6 to 7.2]

5. Secondary Outcome: Physician-reported Ease of Insertion
Description: Measured by VAS (0-100mm; 0 being "very easy", 100 being "very difficult").
Time Frame: Up to 1 minute to complete survey
Population: Participants who received the allocated intervention and for whom primary outcome data are available
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 12 mL Arm | 20 mL Arm
Number analyzed (Participants) | 45 | 46
score on a scale | 27 [13 to 50] | 17 [6 to 28]

6. Secondary Outcome: Count of Participants With Procedural Complications
Time Frame: Up to 10 minutes
Population: Participants who received the allocated intervention and for whom primary outcome data are available
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mL Arm | 20 mL Arm
Number analyzed (Participants) | 45 | 46
Participants | 0 | 0

7. Secondary Outcome: Count of Participants With Side Effects Related to Lidocaine Administration
Description: Side effects were not necessarily considered to be adverse events by investigator.
Time Frame: Up to 10 minutes
Population: Participants who received the allocated intervention and for whom primary outcome data are available
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mL Arm | 20 mL Arm
Number analyzed (Participants) | 45 | 46
Participants
  Metallic taste | 2 | 3
  Ringing in ears | 2 | 3
  Dizziness or lightheadedness | 1 | 6
  Shaky legs | 0 | 1

ADVERSE EVENTS:
Time Frame: Average approximately 45 minutes
Arm/Group | 12 mL Arm | 20 mL Arm
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT03356145/Prot_SAP_001.pdf